CLINICAL TRIAL: NCT00493493
Title: Pore Excision, Curettage, and Injection of a Tissue Scaffold as Treatment for Pilonidal Disease
Brief Title: Pore Excision, Curettage, and Injection of Cymetra for Pilonidal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Matino, James, M.D. (Individual)
Collaborators: LifeCell (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pilonidal/Cymetra
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Pilonidal Sinus
Keywords: Cymetra
MeSH Terms: conditions — Pilonidal Sinus | interventions — Surgical Procedures, Operative; Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: surgery (Pore Excision, Curettage, and Injection of Cymetra)

SUMMARY:
Chronic pilonidal disease is a common problem with no ideal treatment. This is a prospective study that will evaluate the results of surgical pore excision, curettage, and injection of a regenerative tissue matrix, Cymetra, on patients with chronic pilonidal disease.

DETAILED DESCRIPTION:
In addition, the study will evaluate the credibility and reproducibility of results within other surgeons trained to perform the procedure. Data collection will focus on post-operative wound failure, infection ratwes, analgesic requirements, time lost from work or school, wound care requirements, and 6 month recurrence rates. These outcomes will be compared to outcomes using conventional pilonidal surgical intervention using published data.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with pilonidal diseas

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
wound failure, time lost from work or school, analgesic requirements, recurrence rates | 6 months

SECONDARY OUTCOMES:
infection rates, wound care requirements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James J Matino, MD, Principal Investigator — Surgical Group,PC
Locations (1):
- St Francis Hospital, Hartford, Connecticut, United States